CLINICAL TRIAL: NCT06426524
Title: Efficacy of Insulin Like Growth Factor-1(IGF-1) on Bone Regeneration in Intrabony Defects : A Clinico-radiograph Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, PROFFESSOR AND HEAD OF THE DEPARTMENT, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVSInstituteDS1
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Intrabony Periodontal Defect
MeSH Terms: interventions — Durapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): In test group, after reflection of flap and degranulation, IGF-1 gel with hydroxyapatite will be placed in the defect and sutures will be placed.
  Interventions: Procedure: IGF-1 Gel
- Control group (Active Comparator): In control group, after reflection of flap and degranulation, hydroxyapatite will be placed in the defect and sutures will be placed.
  Interventions: Procedure: Hydroxyapatite

INTERVENTIONS:
Procedure: IGF-1 Gel — After degranulation of the defect, IGF-1 gel mixed with Hydroxyapatite graft will be placed in the defect.
  Arms: Test group
Procedure: Hydroxyapatite — After degranulation of the defect, Hydroxyapatite graft will be placed in the defect.
  Arms: Control group

SUMMARY:
The aim of this study is to clinically evaluate the efficacy of Insulin like Growth Factor (IGF-1) on bone regeneration in intrabony defects.

DETAILED DESCRIPTION:
In test group, after reflection of flap and degranulation, IGF-1 gel with hydroxyapatite will be placed in the defect and sutures will be placed.

In control group, after reflection of flap and degranulation, hydroxyapatite will be placed in the defect and sutures will be placed.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy male and female patients of age >18 years Intrabony defects - two wall or three wall defects Probing pocket depths (PPD) of >5mm.

Exclusion Criteria:

Medically compromised patients Pregnant women Heavy smokers Patients who underwent radiotherapy or chemotherapy are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Bone Regeneration | 3 months and 6 months
  Radiovisiography (RVG) will be used to assess bone regeneration achieved post operatively after 3 months and 6 months.
clinical attachment level | 3 months and 6 months
  Assessment of clinical attachment level using UNC-15 probe at baseline and post operatively at 3 and 6 months.
Probig depth | 3 months and 6 months
  Assessment of probing depth using UNC-15 probe at baseline and postoperatively at 3 and 6 months.

SECONDARY OUTCOMES:
Plaque Index | 3 months and 6 months
  Assessment of plaque (PI) - according to Turesky modification of Quigley and Hein Plaque Index, 1970.

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Telangana, India